**Study Protocol – Cover Page** 

Official Study Title:

A Prospective, Randomized Study Comparing the Effect of Alfuzosin, Mirabegron, and Their

Combination on DJ Stent-Related Symptoms After RIRS

NCT Number: (Pending)

Document Type: Study Protocol

Date: May 22, 2025

Sponsor: Gaziantep University

Principal Investigator: Dr. Mehmet Öztürk

COMPARISON OF THE EFFICACY OF ALPHA-BLOCKERS AND

MIIRABEGRON ON SYMPTOMS ASSOCIATED WITH DI STENT

IMPLANTED AFTER RETROGRADE INTRARENAL SURGERY

**ABSTRACT** 

Introduction: This study aimed to evaluate the efficacy of alfuzosin, mirabegron, and their

combination on stone-free rates, residual fragments, stent-related pain, and lower urinary tract

symptoms (LUTS) in patients undergoing double-I (DI) stent placement following retrograde

intrarenal surgery (RIRS).

Methods: A prospective, randomized, single-center trial was conducted between February 2022

and December 2023 at Gaziantep University. A total of 103 patients who underwent RIRS for

unilateral renal stones (1–2 cm) followed by DJ stenting were enrolled. Patients were randomized

into four groups: Group 1 (control, no medication), Group 2 (alfuzosin 10 mg/day), Group 3

(mirabegron 50 mg/day), and Group 4 (alfuzosin + mirabegron). Pain and LUTS were assessed at

30 days postoperatively using the Visual Analog Scale (VAS) and Overactive Bladder-Validated 8

(OAB-V8) form.

Results: The mean age was 43.55 ± 13.93 years. No statistically significant difference was found

between groups in stone-free rates, residual stones, pain, or LUTS (p > 0.05). Group 2 (alfuzosin)

had the lowest mean VAS  $(1.69 \pm 1.52)$  and OAB-V8  $(13.5 \pm 7.37)$  scores, though not statistically

significant when compared to the control group (p = 0.112 and p = 0.592, respectively). Residual stones were detected in 27.2% of patients, and stone size was a significant predictor (p = 0.025).

**Conclusion:** The use of alfuzosin and mirabegron alone or in combination did not have a significant effect on stone-free rates, procedural pain and LUTS. However, alfuzosin may have potential benefits in both pain control and favorable effects on storage symptoms. Further larger-scale studies are warranted.

Keywords: Retrograde intrarenal surgery, double-J stent, alfuzosin, mirabegron, stent-related symptoms